CLINICAL TRIAL: NCT04102891
Title: Health Improvement Through Food and Lifestyle Intervention Based On Personalized Retail Advice
Acronym: FLORA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SmartWithFood (Industry)
Collaborators: Vlaams Instituut voor Biotechnologie (Unknown); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S63023
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome; Gut Bacteria; Personalized Nutrition
Keywords: Metabolic syndrome; Gut microbiota; Personalized dietary advice; Food literacy
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): During the three months intervention period, participants within this arm will do their groceries through the online Collect&Go platform of Colruyt Group. Dietitians will adjust their shopping carts by changing food products by healthier alternative ones taking into account the Flemish food-based dietary guidelines. Based on participants' dietary pattern and level of food literacy, personalized dietary advice will be provided and a dietitian helpline will be available for further nutrition-related questions.
  Interventions: Other: Microbiota modulation diet
- Control arm (No Intervention): During the three months intervention period, participants within this arm will do their groceries through the online Collect&Go platform of Colruyt Group. Dietitians will adjust their shopping carts by changing food products by healthier alternative ones taking into account the guidelines from the newly developed microbiota modulation diet (MMD). Based on participants' dietary pattern and level of food literacy, personalized dietary advice will be provided and a dietitian helpline will be available for further nutrition-related questions.

INTERVENTIONS:
Other: Microbiota modulation diet — The Collect&Go shopping carts of the 400 participants will be adapted by replacing food products by healthier alternative ones based on the Flemish food-based dietary guidelines and the microbiota modulation diet guidelines for the control and study arm respectively. Based on these guidelines, and the habitual dietary pattern and level of food literacy of the participant, personalized dietary advice will be provided. A dietitian helpline will be available for further nutritional issues as well.
  Arms: Study arm

SUMMARY:
FLORA is a longitudinal intervention study with a randomized, parallel group design. Primary objective is to improve metabolic health through gut microbiota modulation by means of a retailer-driven personalized dietary intervention in a real-life setting. Four hundred Flemish pre-metabolic adults will be randomly divided into a control and treatment arm, each comprising 200 participants. The study period is divided into three phases: a four weeks characterization, a twelve weeks intervention, and a four weeks post-intervention phase. During the intervention phase, control participants' online Collect&Go shopping carts are adjusted in accordance with Flemish food-based dietary guidelines. Based on the same guidelines, participants are provided with personalized dietary advice considering their usual dietary pattern and level of food literacy. In the treatment arm, a similar intervention will be applied using guidelines based on a microbiota modulation diet (MMD). During intervention, all participants can contact a dietician helpline for additional advice on study-related dietary issues. Over the five months, saliva and fecal samples will be collected on a regular basis, with an intensive sampling period of seven consecutive days at the end of each study phase. A GP consult consisting of a short medical exam, blood withdrawal and medical questionnaire takes place each month. Further, online questionnaires on lifestyle, health and well-being will be sent by e-mail and each five days, participants complete a food diary through their smartphone. Fecal, saliva, blood samples and meta-data will be analysed to detect changes in metabolic health.

ELIGIBILITY:
Inclusion criteria

* Willingness to participate to the study and to sign the informed consent (Dutch)
* Older than 18 years
* Diagnosed with pre-metabolic syndrome (diagnosed with central obesity [waist circumference ≥80 cm for women and ≥94 cm for men] and one of the following criteria: elevated blood pressure [systolic ≥130 mm Hg, diastolic ≥85 mm Hg], raised triglycerides [>150 mg/dL], reduced HDL-cholesterol [<40 mg/dL in men, <50 mg/dL in women], or raised fasting plasma glucose [≥100 mg/dL]
* Residing in Belgium, no travels abroad planned longer than seven consecutive days during the five-months study period
* Willingness to follow dietary guidelines during the three-months intervention period
* Willingness to purchase bulk groceries primarily at Colruyt Group using the Collect&Go platform during the five-months study period
* Access to a -20-18°C freezer

Exclusion criteria

* Chronic constipation (less than one defecation once a week)
* Gastro-intestinal surgery within the past 3 months
* Inflammatory bowel disease (IBD) or diverticulitis
* Irritable bowel syndrome (IBS)
* Any food allergy or food intolerance
* Metabolic syndrome
* Diabetes Mellitus Type 1 or Type 2
* Coeliac disease
* Pregnant women or women planning a pregnancy during the study period
* Lactating women
* Subjects on a specific diet (e.g. vegetarian/vegan diet, gluten-free diet, lactose-free diet, high-protein diet)
* Subjects being treated for hypertension or high cholesterol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Reduced waist circumference | 5 months
  Participants' waist circumference (cm) decreases during the study period
Reduced serum triglycerides | 5 months
  Participants' serum triglyceride level (mg/dL) decreases during the study period (blood sample analysis)
Reduced blood pressure | 5 months
  Participants' blood pressure (mm Hg) decreases during the study period
Elevated HDL-cholesterol | 5 months
  Participants' HDL-cholesterol levels (mg/dL) increase during the study period (blood sample analysis)
Reduced fasting plasma glucose | 5 months
  Participants' fasting plasma glucose levels decrease during the study period (blood sample analysis)

IPD SHARING:
Plan to Share IPD: No